CLINICAL TRIAL: NCT00530569
Title: Evaluation of Clinical Significance of Circulating Markers in Breast Cancer Patients Undergoing Herceptin Therapy
Acronym: HER 2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: 17924
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Herceptin Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood Test — CBC and HER2 level at baseline, prior to each chemo and/or herceptin cycle, one month after chemo and/or herceptin completion, quarterly up to 12 months or a maximum of 20 blood draws.

SUMMARY:
About 30% of breast cancers have higher than normal levels of a cellular marker called HER2. The amount of HER2 is often measured in breast tissue. A higher level of this marker usually indicates a more aggressive type of breast cancer. Cytokeratin is a second cellular marker found in breast cancer cells. Detection of Circulating cytokeratin in the blood could indicate the presence of cancer. The Pathology Department of the Tom Baker Cancer Center is doing this study to see if measuring the levels of circulating HER2 and cytokeratin, through blood testing has clinical significance for patients with breast cancer.

DETAILED DESCRIPTION:
* Single Variate analysis will be performed to correlate variables such as tumour size, grade, stage, ER status, PR status and biopsy HER2 status with soluble HER2 levels.
* Soluble HER2 levels will be analyzed as both a continuous and categorized variable.
* The analysis will attempt to discern the relationship between soluble HER2 levels, HER2 positive circulating epithelial cell level and treatment response.
* This will provide evidence of the effect various treatments have on HER2 levels. HER2 levels both in patients treated with Herceptin and those on other treatment protocols, will be related to clinical disease measures such as time to progression, time to failure, duration of response and duration of survival.
* An initial model of the relationship between these factors and soluble HER2 as a marker will be established from the data.

ELIGIBILITY:
Inclusion Criteria:

* Albertan women with breast cancer who will undergo Herceptin therapy as part of their treatment at some point during a one-year period.

Exclusion Criteria:

* Greater than 80 years of age
* Previous cancer diagnosis - (other than skin cancer)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Albertan women with breast cancer who will undergo Herceptin therapy as part of their treatment at some point during a one-year period.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Bill Kangerloo, M.D., Principal Investigator — Alberta Health services
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada